CLINICAL TRIAL: NCT02913040
Title: High Flow Nasal Cannula Therapy for Infants With Bronchiolitis
Brief Title: High Flow in Infants With Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Amalia Children's Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: High Flow in Bronchiolitis
Record Dates: First submitted 2016-09-17; First posted 2016-09-23 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Flow Nasal Cannula (Experimental): Oxygen delivery through Heated Humidified High Flow Nasal Cannula
  Interventions: Other: High Flow Nasal Cannula
- Low Flow Nasal Prongs (Active Comparator): Oxygen delivery through Low Flow Nasal Prongs
  Interventions: Other: Low Flow Nasal Prongs

INTERVENTIONS:
Other: High Flow Nasal Cannula — Oxygen delivery through Heated Humidified High Flow Nasal Cannula
  Other Names: HFNC
  Arms: High Flow Nasal Cannula
Other: Low Flow Nasal Prongs — Oxygen delivery through Low Flow Nasal Prongs
  Other Names: LFNC
  Arms: Low Flow Nasal Prongs

SUMMARY:
In this multi-centre randomized controlled trial the investigators compare the effect on dyspnoea severity of oxgen delivery through High Flow Nasal cannula with Low Flow Nasal Prongs in children < 2 years of age hospitalised for bronchiolitis with moderate-severe dyspnoea.

DETAILED DESCRIPTION:
In this multi-centre randomized controlled trial the investigators compare the effect on dyspnoea severity of oxgen delivery through High Flow Nasal Cannula with Low Flow Nasal Prongs in children < 2 years of age hospitalised for bronchiolitis with moderate-severe dyspnoea. The study will take place on the pediatric (Non intensive care) units of 5 different hospitals in the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* bronchiolitis PEWS (Pediatric Early Warning Score 0-28) >= 6 oxygen saturation < 92%

Exclusion Criteria:

* chronic lung disease hemodynamic significant heart disease syndromal disease facial abnormalities

Ages: 1 Week to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
PEWS (Pediatric Early Warning Score) (in points 0-28) | 24 hours
  Sustained reduction in PEWS >= 2 points within 24 hours (min 0- max 28 points)

SECONDARY OUTCOMES:
Comfort (in points 0-10) | 24 hours
  (FLACC: Face, Legs, Activity, Cry, Consolability, min 0- max 10 points)
ability to feed (yes or no) | 5 days
  need for tubefeeding and/or intravenous fluids
duration of hospitalisation in days | 15 days
  duration of hospitalisation in days
admission to PICU (Pediatric Intensive Care Unit) (yes or no) | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Jolita Bekhof, MD, PhD, Principal Investigator — Isala
Locations (7):
- Netherlands (7):
  - Isala Klinieken, Zwolle, Overijssel
  - Amphia, Breda
  - Deventer Ziekenhuis, Deventer
  - Medisch Spectrum Twente, Enschede
  - Martini Ziekenhuis, Groningen
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - Ikazia Hospital, Rotterdam

IPD SHARING:
Plan to Share IPD: Yes
publication in journal
Supporting Information: Study Protocol, CSR
Time Frame: after publication in a journal

REFERENCES:
- [Derived] Kooiman L, Blankespoor F, Hofman R, Kamps A, Gorissen M, Vaessen-Verberne A, Heuts I, Bekhof J. High-flow oxygen therapy in moderate to severe bronchiolitis: a randomised controlled trial. Arch Dis Child. 2023 Jun;108(6):455-460. doi: 10.1136/archdischild-2022-324697. Epub 2023 Mar 20. PMID 36941030